CLINICAL TRIAL: NCT02863380
Title: Validation of Personalized Antidepressant Treatment by Neuromodulation - Pilot Study
Brief Title: Personalized rTMS for Resistant Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The research objectives are achieved, demonstrating the feasibility and superiority of the personalized approach. It was no longer justified to continue the inclusions in this 'proof of concept' type study.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 6194
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder; Treatment-Resistant
Keywords: Individualized Medicine; Transcranial Magnetic Stimulation, Repetitive; Transcranial Direct Current Stimulation Monocentric; Compariative Cross-Over 3 Arms Study Randomized, Single-Blind Method; Functional Neuroimaging
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individualized rTMS (transcranial magnetic stimulation) (Experimental): The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 38). rCBF will be measured using the QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio.
  The therapeutic protocol will be design to correct the rCBF anomaly first by defining each point where to deliver the stimulation than the stimulation protocol for each point (180% of active motor threshold, 4-second 10 Hz train duration, with 26-second intertrain interval for a total of 3000 pulses). The whole target will be homogeneously stimulated.
  The active motor threshold will be assessed. The procedure will be repeated twice a day for 10 days over 2 weeks.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol; Device: Individualized rTMS (transcranial magnetic stimulation)
- Classical rTMS (transcranial magnetic stimulation) (Active Comparator): rTMS will be performed as usual using a figure-eight coil: Defining the active motor threshold. For each session positioning the coil on F3, stimulating at 180% of active motor threshold (10 Hz, 4-second train duration, and 26-second intertrain interval) for 37.5 minutes (3000 pulses per session), twice a day for 10 days over 2 weeks.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol; Device: Classical rTMS (transcranial magnetic stimulation)
- Classical tDCS (transcranial direct current stimulation) (Active Comparator): tDCS will be performed as usual: After controlling for skin healthiness, the anode and the cathode will be respectively placed over F3 and right shoulder. A commercial devices (MagStim), will deliver a constant current of 2 mA through 25 cm2 saline-soaked rubber sponges for 20 min per session. The procedure will be repeated twice a day for 10 days over 2 weeks.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol; Device: Classical tDCS (transcranial direct current stimulation)

INTERVENTIONS:
Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol — Procedure consisting in personalizing the rTMS targets and stimulation pattern based on functional magnetic resonance imaging
Device: Individualized rTMS (transcranial magnetic stimulation)
  Arms: Individualized rTMS (transcranial magnetic stimulation)
Device: Classical rTMS (transcranial magnetic stimulation)
  Arms: Classical rTMS (transcranial magnetic stimulation)
Device: Classical tDCS (transcranial direct current stimulation)
  Arms: Classical tDCS (transcranial direct current stimulation)

SUMMARY:
The investigators hypothesize that personalizing the rTMS targets using functional MRI will increase its efficacy. The most dysfunctional regions or the most dysfunctional network will be stimulated homogeneously. Individualized rTMS will be compared to traditional rTMS procedure and to trans-cranial direct current stimulation (tDCS) in a randomized cross-over trial.

In this pilot study the primary outcome measure will be the correction of the MRI anomalies. Symptoms reduction and the proportion of remitters will be secondary outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 Y
* Affiliated to the health insurance
* Having signed an informed consent
* Suffering from major depression according to the DSM5
* Unresponsive or incomplete remission after at least one trial of antidepressant (> 6 weeks at efficient dose or side effects)
* Treatment stable for > 6 weeks

Exclusion Criteria:

* Contraindication for MRI, rTMS or tDCS: non-removable ferromagnetic body, prosthesis, pacemaker, medication delivered by an implanted pump clip or vascular stent, heart valve or ventricular shunt, seizure disorders, skin pathology in the region of tDCS electrode placement.
* Pregnancy
* Severe and non-stabilized somatic pathology
* Patients deprived of liberty or hospitalized without their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Change of rCBF anomalies | Difference between before (assessed once between D-7 to -1) and after (assessed once between D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  The target region will be defined by comparing the rCBF scan of the patient to a control population. rCBF will be measured using the average of 2 ∙ 3 (=6) measures of rCBF using QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio. rCBF change of the target region will be compared before & after therapeutic protocol between the different procedures (ANOVA).
  Functional connectivity map of the target region will be performed by extracting its average temporal course and looking at the region(s) which activity is correlated. Contrast map of each patient will be compared to the one of a control population submitted to the same analysis. Change in the number of above threshold voxels (F-test, p < 0.05 uncorrected, extension > 1 cm3) will be compared before & after therapeutic procedure (ANOVA). rCBF's change of the target region will be compared before & after therapeutic protocol between the different procedures (ANOVA).
Change of the functional connectivity anomalies | Difference between before (assessed once between D-7 to -1) and after (assessed once between D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  The target region will be defined by comparing the rCBF scan of the patient to a control population. rCBF will be measured using the average of 2 ∙ 3 (=6) measures of rCBF using QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio. rCBF change of the target region will be compared before & after therapeutic protocol between the different procedures (ANOVA).
  Functional connectivity map of the target region will be performed by extracting its average temporal course and looking at the region(s) which activity is correlated. Contrast map of each patient will be compared to the one of a control population submitted to the same analysis. Change in the number of above threshold voxels (F-test, p < 0.05 uncorrected, extension > 1 cm3) will be compared before & after therapeutic procedure (ANOVA). rCBF's change of the target region will be compared before & after therapeutic protocol between the different procedures (ANOVA).

SECONDARY OUTCOMES:
Change in symptoms evaluated by the clinician (QIDS16-C) | Difference between before (assessed once between D-7 to -1) and after (assessed once between D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
  See http://www.ids-qids.org/ for documentation relative to these scales. Computation will be performed in terms of : percentage of symptom reduction Number responders (reduction of more than 50% of symptoms) & numbers of remitters (QIDS16-C ≤ 6).
Change in symptoms evaluated by the patient (QIDS30-SR) | Difference between before (assessed once between D-7 to -1) and after (assessed once between D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
  See http://www.ids-qids.org/ for documentation relative to these scales. Computation will be performed in terms of : percentage of symptom reduction Number responders (reduction of more than 50% of symptoms) & numbers of remitters (QIDS16-C ≤ 6).

OTHER OUTCOMES:
Daily visual analogical scales assessing the core symptoms | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
Response time and accuracy at the attentional network test | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
Quality of life ("Echele synoptique des 3 temps") | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
Global Assessment of Functioning | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Jack FOUCHER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Psychiatrie 1, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dormegny-Jeanjean LC, de Crespin de Billy C, Pierrat C, Mainberger O, Schorr B, Obrecht A, Arcay H, Moreau A, Humbert I, Scarlatti F, Bertschy G, de Sousa PL, Lamy J, Weibel S, Landre L, Foucher JR. Individualizing rTMS in treatment-resistant depression from patient-specific perfusion abnormalities a proof-of-concept randomized trial in comparison to standard rTMS and tDCS. Eur Arch Psychiatry Clin Neurosci. 2025 Sep;275(6):1809-1825. doi: 10.1007/s00406-025-02027-7. Epub 2025 Jun 14. PMID 40517147